CLINICAL TRIAL: NCT05785793
Title: Clinical Characteristics and Outcomes of Autoimmune Hepatitis: a Retro-prospective Multicenter Cohort in China
Brief Title: Autoimmune Hepatitis Cohort in China
Acronym: CAMERA
Status: Recruiting | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, maxiong, Director of Gastroenterology and Hepatology, Renji Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: AIH-CH
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Autoimmune Hepatitis
MeSH Terms: conditions — Hepatitis, Autoimmune

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — blood samples and liver biopsy specimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to describe the clinical features and long-term prognosis in patients diagnosed with autoimmune hepatitis (AIH) in China and assess the effectiveness and safety of AIH treatment options in a real-world setting.

DETAILED DESCRIPTION:
Autoimmune hepatitis (AIH) is a chronic autoimmune liver disease that causes liver inflammation and necrosis, ultimately leading to cirrhosis and liver failure. Although relatively rare, the prevalence of AIH in China has been increasing in recent years, highlighting its significance as a public health issue. However, due to the wide variability in the clinical presentation and outcomes of AIH, diagnosing and managing the disease can be challenging. Moreover, our understanding of the epidemiology, clinical features, diagnosis, and treatment of AIH in China is still limited.

To address this gap in knowledge, the investigators are conducting the Chinese AIH Cohort study, which collects data from approximately 20 sites across China on treatment progress and success in clinical routine. The study aims to evaluate the effectiveness and safety/tolerability of different AIH treatment options, including standard therapy, and second and third-line treatment options. The investigators also record the long-term prognosis of patients with AIH, tracking whether they achieve remission, require liver transplantation, or experience mortality. Risk factors associated with long-term prognosis and survival will be analyzed to provide insights that can improve the diagnosis, treatment, and management of AIH in this population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 14 years
* Probable or definite diagnosis of autoimmune hepatitis according to the International Autoimmune Hepatitis Study Group criteria
* Availability of all following essential parameters at the initial diagnosis of AIH: including alanine transaminase, aspartate aminotransferase, total bilirubin, alkaline phosphatase, immunoglobulin G, and platelet count
* Provide informed consent

Exclusion Criteria:

* Have a concomitant diagnosis of primary biliary sclerosis, primary sclerosing cholangitis, immunoglobulin G 4-related cholangitis
* Have an active infection with hepatitis B virus, hepatitis C virus, hepatitis delta virus, HIV, cytomegalovirus, or Epstein-Barr virus
* Have a concomitant diagnosis of hepatocellular carcinoma or other malignant diseases before the diagnosis of AIH
* Considered ineligible to the enrollment in the clinical study by the researcher

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients diagnosed as AIH in medical centers and outpatient clinics.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Transplant free survival | From baseline to 60 months after baseline
  Time to the first occurrence of liver transplant or death from any cause

SECONDARY OUTCOMES:
Liver-related death | From baseline to 60 months after baseline
  Time to the first occurrence of liver transplant or death from liver-related cause
Biochemical response | From baseline to 60 months after baseline
  Proportion of patients who achieve complete biochemical response (normalisation of serum transaminases and immunoglobulin G below the ULN)
Remission | From baseline to 60 months after baseline
  Proportion of patients who achieve remission (hepatitis activity index<4/18)
Complications | From baseline to 60 months after baseline
  Occurrence of variceal hemorrhage, ascites, jaundice, encephalopathy and hepatocellular carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Xiong Ma, MD,PHD, Study Chair — Renji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China